CLINICAL TRIAL: NCT00700791
Title: Efficacy of Natural Vitamin E Tocotrienol on the Treatment of Surgical Scars
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The PI moved to another Institution
Sponsor: Chandan K Sen (Other)
Responsible Party: Sponsor-Investigator, Chandan K Sen, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2008H0001
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Scar
Keywords: Single and bilateral body contouring surgical sites.
MeSH Terms: conditions — Cicatrix | interventions — Thrombin Time

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Group I Single Site Randomization (Placebo Comparator): Patients with 1 surgical scar will be given both oral placebo and topical cream placebo
  Interventions: Other: Placebo; Other: Placebo Cream
- Group II Single Site Randomization (Active Comparator): Single surgical site will be given oral placebo and topical TCT
  Interventions: Device: Natural Vitamin E Tocotrienol Cream (TCT); Other: Placebo
- Group III Single Site Randomization (Active Comparator): Patients with 1 surgical scar will be given Natural Vitamin E Tocotrienol supplement (TCT) and topical placebo cream
  Interventions: Dietary Supplement: Natural Vitamin E Tocotrienol supplement (TCT); Other: Placebo Cream
- Group IV Single Site Randomization (Active Comparator): Patients with 1 surgical scar will be given both Natural Vitamin E Tocotrienol supplement (TCT) and Natural Vitamin E Tocotrienol Cream (TCT).
  Interventions: Dietary Supplement: Natural Vitamin E Tocotrienol supplement (TCT); Device: Natural Vitamin E Tocotrienol Cream (TCT)
- Group I: Bilateral Site Randomization (Placebo Comparator): Patients with bilateral surgical scars will be given both oral placebo and topical cream placebo on one surgical site.
  Interventions: Other: Placebo; Other: Placebo Cream
- Group II: Bilateral Site Randomization (Active Comparator): Patients with bilateral surgical scars will be given oral placebo and Natural Vitamin E Tocotrienol Cream (TCT) to one of the surgical sites.
  Interventions: Device: Natural Vitamin E Tocotrienol Cream (TCT); Other: Placebo
- Group III: Bilateral Site Randomization (Active Comparator): Patients with bilateral surgical scars will be given Natural Vitamin E Tocotrienol supplement (TCT) and topical placebo cream on one surgical site.
  Interventions: Dietary Supplement: Natural Vitamin E Tocotrienol supplement (TCT); Other: Placebo Cream
- Group IV: Bilateral Site Randomization (Active Comparator): Patients with bilateral surgical scars will be given Natural Vitamin E Tocotrienol supplement (TCT) and Natural Vitamin E Tocotrienol Cream (TCT) on one surgical site.
  Interventions: Dietary Supplement: Natural Vitamin E Tocotrienol supplement (TCT); Device: Natural Vitamin E Tocotrienol Cream (TCT)
- Normal Skin and Adipost Tissue Group (No Intervention): Normal human skin and adipose tissue will be collected

INTERVENTIONS:
Dietary Supplement: Natural Vitamin E Tocotrienol supplement (TCT) — Oral Vitamin E Tocotrienol Supplement (TCT)
  Other Names: Oral TCT
  Arms: Group III Single Site Randomization; Group III: Bilateral Site Randomization; Group IV Single Site Randomization; Group IV: Bilateral Site Randomization
Device: Natural Vitamin E Tocotrienol Cream (TCT) — Natural Vitamin E Tocotrienol(TCT)Topical Cream
  Other Names: Topical TCT
  Arms: Group II Single Site Randomization; Group II: Bilateral Site Randomization; Group IV Single Site Randomization; Group IV: Bilateral Site Randomization
Other: Placebo — Oral Placebo
  Arms: Group I Single Site Randomization; Group I: Bilateral Site Randomization; Group II Single Site Randomization; Group II: Bilateral Site Randomization
Other: Placebo Cream — Topical Placebo Cream
  Arms: Group I Single Site Randomization; Group I: Bilateral Site Randomization; Group III Single Site Randomization; Group III: Bilateral Site Randomization

SUMMARY:
The overall goal of this study is to determine the efficacy of tocotrienol (TCT), a natural form of vitamin E, in preventing or reducing scar formation in human skin wounds as well as the basal levels of TCT in normal human skin and adipose tissue.

DETAILED DESCRIPTION:
Scar formation is the physiological and inevitable end point of mammalian wound healing and there is substantial evidence that inflammation is an essential prerequisite for scarring. Although scar tissue restores the normal skin barrier, the new tissue is inferior in structural, aesthetic, and functional respects. The mammalian wound healing response may have originated during the time of high susceptibility to infection. Therefore, we may have developed speed optimized wound healing where a multiple redundant compensating rapid inflammatory response allows the wound to heal quickly without infection. The scar is then the price mammals have to pay for evolutionary survival after being wounded.

Tocotrienol may be an effective tool to prevent or reduce normal, hypertrophic, or keloid scarring by mediating the inflammatory response. Tocotrienol is a safe and convenient treatment that could be used by mouth or topically. There has never been a study on the effectiveness of tocotrienol in preventing or reducing scar formation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Non- smoker
* No current medications that alter liver metabolism (e.g., Phenobarbital, HmG co-A inhibitors, etc.)
* Non- pregnant or non-breastfeeding
* No current use of dietary supplements containing vitamin-E
* Not actively abusing drugs or alcohol

Exclusion Criteria:

* Under 18 years of age
* Prisoners
* Current smoker
* Pregnant or breastfeeding
* HIV diagnosis
* Viral hepatitis diagnosis
* Immunosuppressive therapy
* Actively abusing drugs or alcohol
* Current use of dietary supplements containing vitamin-E

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2008-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
1.To determine the efficacy of TCT in improving the appearance of post-surgical scars following oral supplementation 2.To determine the efficacy of TCT in improving the appearance of post-surgical scars following topical application | 4 weeks prior to surgery and 12 weeks post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - OSU Plastic Surgery - Knightsbridge, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio